CLINICAL TRIAL: NCT06934642
Title: Effect of Tirzepatide on Markers of MASLD in Patients With Obesity: A Pilot Study
Brief Title: Effect of Tirzepatide on Markers of MASLD in Patients With Obesity
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: American Cancer Society, Inc. (Other); University of New Mexico Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 25-072
Record Dates: First submitted 2025-04-11; First posted 2025-04-18 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: MASLD; Obesity
MeSH Terms: conditions — Obesity | interventions — Tirzepatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Intervention Arm (Experimental): Individuals in the intervention arm (only arm) will receive tirzepatide for 12 months.
  Interventions: Drug: Tirzepatide

INTERVENTIONS:
Drug: Tirzepatide — The drug is being studied to better understand the biological effects of tirzepatide on MASLD.
  Other Names: Zepbound; Mounjaro

SUMMARY:
Metabolic Dysfunction-Associated Steatotic Liver Disease (MASLD) is the most common cause of chronic liver disease worldwide and predominately affects individuals with overweight and obesity, as well as those with type 2 diabetes and cardiovascular disease. Tirzepatide is a medication used to treat type 2 diabetes and obesity. It has also been shown to help with MASLD. The purpose of this study is to study how tirzepatide affects the liver in patients with MASLD.

Participants will be asked to:

* Take tirzepatide for 12 months.
* Come in for clinic visits every 3 months.
* Have blood drawn at baseline, 6, and 12 months.
* Complete a liver ultrasound at baseline and at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Age 18-75
* Diagnosis of MASLD based on the following criteria:

  * Presence of at least 1 out of the 5 following cardiometabolic criteria:
* BMI >25 kg/m2 OR waist circumference >94 cm (men) or 80cm (women)
* Fasting serum glucose >100 mg/dL OR 2-hour post-prandial glucose levels >140mg/dL OR AbA1c >5.7% OR type 2 diabetes OR treatment for type 2 diabetes
* Blood pressure >130/85 mmHg OR specific antihypertensive drug treatment
* Plasma triglycerides >150mg/dL OR on lipid lowering treatment
* Plasma HDL-cholesterol <40mg/dL (men) and <50mg/dL (women) OR on lipid lowering medication

  * No other identified causes of steatosis
  * Evidence of steatotic liver disease (hepatic steatosis identified by imaging or biopsy)
* English speaking

Exclusion Criteria:

* Pregnancy or breast feeding
* Premenopausal women not on any form of contraception
* Reports alcohol intake >50g/day or 350g/week for women and >60g/day or 420g/week for men or an AUDIT score >8
* Other identifiable causes of steatosis
* Documented allergic reaction to tirzepatide or any other GLP1 RA
* Decompensated liver disease
* Decompensated renal disease requiring hemodialysis
* Decompensated heart failure
* Active malignancy
* Prior history of pancreatitis
* Serum triglyceride levels >500 mg/dL
* Personal or family history of medullary thyroid cancer or MEN2a or MEN2b
* Concurrent use of other ant-obesity medications
* Use of other GLP1 RAs within 3 months of study enrollment
* Unable to obtain the medication due to cost or insurance coverage restrictions.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Biomarkers associated with MASLD | 12 months
  Identification of an changes in biomarkers associated with MASLD with tirzepatide use

SECONDARY OUTCOMES:
Liver Fat Content | 12 months
  Change in liver fat content with use of tirzepatide
Liver Stiffness | 12 months
  Change in liver stiffness with use of tirzepatide
Body weight | 12 months
  Change in body weight with use of tirzepatide
Metabolic markers | 12 months
  Changes in lipid profiles, glycemic measures (A1c), inflammatory markers and cytokines, and gut hormones

CONTACTS AND LOCATIONS:
Overall Officials: Eliseo Castillo, Principal Investigator — UNM Cancer Center
Locations (1):
- University of New Mexico Health Sciences Center, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers. Data will only be available to study team members.